CLINICAL TRIAL: NCT03399448
Title: Phase 1 Trial of Autologous T Cells Engineered to Express NY-ESO-1 TCR and CRISPR Gene Edited to Eliminate Endogenous TCR and PD-1 (NYCE T Cells)
Brief Title: NY-ESO-1-redirected CRISPR (TCRendo and PD1) Edited T Cells (NYCE T Cells)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor has terminated trial to pursue other targets.
Sponsor: University of Pennsylvania (Other)
Collaborators: Parker Institute for Cancer Immunotherapy (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UPCC# 25416; IRB #826672
Record Dates: First submitted 2017-12-20; First posted 2018-01-16 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma; Melanoma; Synovial Sarcoma; Myxoid/Round Cell Liposarcoma
MeSH Terms: conditions — Multiple Myeloma; Melanoma; Sarcoma, Synovial; Liposarcoma, Myxoid | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Multiple Myeloma (MM) (Experimental)
  Interventions: Biological: NY-ESO-1 redirected autologous T cells with CRISPR edited endogenous TCR and PD-1; Drug: Cyclophosphamide; Drug: Fludarabine; Device: NY-ESO-1 expression testing
- Synovial Sarcoma (SS) and Myxoid/Round Cell Liposarcoma (MRCL) (Experimental)
  Interventions: Biological: NY-ESO-1 redirected autologous T cells with CRISPR edited endogenous TCR and PD-1; Drug: Cyclophosphamide; Drug: Fludarabine; Device: NY-ESO-1 expression testing
- Melanoma (Experimental): Not Recruiting at the UPenn Site
  Interventions: Biological: NY-ESO-1 redirected autologous T cells with CRISPR edited endogenous TCR and PD-1; Drug: Cyclophosphamide; Drug: Fludarabine; Device: NY-ESO-1 expression testing

INTERVENTIONS:
Biological: NY-ESO-1 redirected autologous T cells with CRISPR edited endogenous TCR and PD-1 — Autologous T cells transduced with a lentiviral vector to express NY-ESO-1 and electroporated with CRISPR guide RNA to disrupt expression of endogenous TCRα, TCRβ and PD-1 (NYCE T Cells).
Drug: Cyclophosphamide — a cytotoxic chemotherapy agent used for lymphodepletion prior to NYCE T cells.
Drug: Fludarabine — a chemotherapy agent used for lymphodepletion prior to NYCE T cells.
Device: NY-ESO-1 expression testing — Testing to determine if NY-ESO-1 is expressed on tumor tissue.

SUMMARY:
This is a first-in-human trial proposed to test HLA-A*0201 restricted NY-ESO-1 redirected T cells with edited endogenous T cell receptor and PD-1.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a confirmed diagnosis of relapsed refractory multiple myeloma (MM), melanoma, synovial sarcoma, or myxoid/round cell liposarcoma (MRCL) as follows:

a. Multiple Myeloma i. Subjects must have a confirmed prior diagnosis of active MM as defined by the International Myeloma Working Group (IMWG) criteria.

ii. Subjects must have relapsed or refractory disease after either one of the following:

1. At least 3 prior regimens, which must have contained an alkylating agent, proteasome inhibitor, and immunomodulatory agent (IMiD) OR
2. At least 2 prior regimens if "double-refractory" to a proteasome inhibitor and IMiD, defined as progression on or within 60 days of treatment with these agents.

Note: Induction therapy, stem cell transplant, and maintenance therapy, if given sequentially without intervening progression, should be considered as 1 "regimen".

iii. Subjects must be at least 90 days since autologous stem cell transplant, if performed.

iv. Toxicities from prior therapies, with the exception of alopecia or peripheral neuropathy attributable to bortezomib, must have recovered to grade ≤ 2 according to the Common Toxicity Criteria (CTCAE) 4.0 criteria or to the subject's prior baseline.

v. Subjects must have measurable disease per IMWG criteria on study entry, which must include at least 1 of the following:

1. Serum M-spike ≥ 0.5 g/dL*
2. 24 hour (hr) urine M-spike ≥ 200mg
3. Involved serum free light chain (FLC) ≥ 50 mg/L with abnormal ratio
4. Measurable plasmacytoma on exam or imaging
5. Bone marrow plasma cells ≥ 20%

   * Note: Patients with IgA myeloma in whom serum protein electrophoresis is deemed unreliable, due to co-migration of normal serum proteins with the paraprotein in the beta region, may be considered eligible as long as total serum IgA level is elevated above normal range.

     b. Melanoma i. Subjects must have a confirmed prior diagnosis of melanoma. ii. Progressed after at least 2 therapy lines. iii. Subjects with BRAF mutant tumors should have received and progressed through, or are intolerant to, BRAF/MEK inhibitor therapy prior to enrollment iv. Patients must have measurable disease per RECIST 1.1 in order to allow assessment of an anti-tumor response.

     c. Synovial Sarcoma or Myxoid/Round Cell Liposarcoma (MRCL) i. Subjects must have a confirmed prior diagnosis of synovial sarcoma or MRCL. ii. Patients with proven metastatic disease or surgically inoperable local recurrence that have failed first line treatment.

iii. Patients must have measurable disease per RECIST 1.1 in order to allow assessment of an anti-tumor response.

2. Provides written, informed consent. 3. Subjects ≥ 18 years of age. 4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. 5. Documented NY-ESO-1 and/or LAGE-1 expression on tumor tissue. 6. HLA-A*201 positive 7. Subjects of reproductive potential must agree to use acceptable birth control methods.

8. Adequate vital organ function as defined by:

1. Serum creatinine ≤ 2.5 or estimated creatinine clearance ≥30 ml/min and not dialysis-dependent.
2. Absolute neutrophil count ≥1000/μl and platelet count ≥50,000/μl (≥30,000/μl if bone marrow plasma cells are ≥50% of cellularity for MM patients).
3. Serum glutamic oxaloacetic transaminase (SGOT) ≤ 3x the upper limit of normal and total bilirubin ≤ 2.0 mg/dl (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome).
4. Left ventricular ejection fraction (LVEF) ≥ 45%. LVEF assessment must have been performed within 8 weeks of eligibility confirmation by physician-investigator.

Exclusion Criteria:

* 1. Pregnant or nursing (lactating) women.
* 2. Have inadequate venous access for or contraindications to leukapheresis.
* 3. Have any active and uncontrolled infection.
* 4. Active hepatitis B or hepatitis C
* 5. Human immunodeficiency virus (HIV) infection.
* 6. Any uncontrolled medical or psychiatric disorder that would preclude participation as outlined.
* 7. New York Heart Association (NYHA) Class III or IV heart failure, unstable angina, or a history of recent (within 6 months) myocardial infarction or sustained (>30 seconds) ventricular tachyarrhythmias.
* 8. Received prior gene therapy or gene-modified cellular immunotherapy. Subject may have received, however, non-gene-modified autologous T-cells in association with an anti-myeloma vaccine (e.g., hTERT or MAGEA3) or vaccination against infectious agents (e.g., influenza or pneumococcus) as was performed on our previous studies.
* 9. Active auto-immune disease, including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis, or have a history of severe (as judged by the principal investigator) autoimmune disease requiring prolonged immunosuppressive therapy.
* 10. Prior allogeneic stem cell transplant.
* 11. Prior or active central nervous system (CNS) involvement (e.g. leptomeningeal disease, parenchymal masses) with myeloma. Screening for this (e.g. with lumbar puncture) is not required unless suspicious symptoms or radiographic findings are present. Subjects with calvarial disease that extends intracranially and involves the dura will be excluded, even if cerebrospinal fluid (CSF) is negative for myeloma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Determine safety profile of a single infusion of NYCE T cells by monitoring the frequency and severity of adverse events assessed by the National Cancer Institute (NCI) - Common Toxicity Criteria (v4.03) | 5 years
Evaluate Manufacturing Feasibility of NYCE T Cells. | 5 years
  Evaluate the percentage of manufacturing products that do not meet release criteria for vector transduction efficiency, gene disruption T cell product purity, viability, sterility or due to tumor contamination.

SECONDARY OUTCOMES:
Percentage of patients achieving complete response (CR) before or at Month 6 | 6 months
Overall survival (OS) | 5 years
Duration of remission (DOR) | 5 years
Progression- free survival (PFS) | 5 years
Cause of death (COD) when appropriate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward Stadtmauer, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stadtmauer EA, Fraietta JA, Davis MM, Cohen AD, Weber KL, Lancaster E, Mangan PA, Kulikovskaya I, Gupta M, Chen F, Tian L, Gonzalez VE, Xu J, Jung IY, Melenhorst JJ, Plesa G, Shea J, Matlawski T, Cervini A, Gaymon AL, Desjardins S, Lamontagne A, Salas-Mckee J, Fesnak A, Siegel DL, Levine BL, Jadlowsky JK, Young RM, Chew A, Hwang WT, Hexner EO, Carreno BM, Nobles CL, Bushman FD, Parker KR, Qi Y, Satpathy AT, Chang HY, Zhao Y, Lacey SF, June CH. CRISPR-engineered T cells in patients with refractory cancer. Science. 2020 Feb 28;367(6481):eaba7365. doi: 10.1126/science.aba7365. Epub 2020 Feb 6. PMID 32029687
- [Derived] Tsuchida CA, Brandes N, Bueno R, Trinidad M, Mazumder T, Yu B, Hwang B, Chang C, Liu J, Sun Y, Hopkins CR, Parker KR, Qi Y, Hofman L, Satpathy AT, Stadtmauer EA, Cate JHD, Eyquem J, Fraietta JA, June CH, Chang HY, Ye CJ, Doudna JA. Mitigation of chromosome loss in clinical CRISPR-Cas9-engineered T cells. Cell. 2023 Oct 12;186(21):4567-4582.e20. doi: 10.1016/j.cell.2023.08.041. Epub 2023 Oct 3. PMID 37794590
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818